CLINICAL TRIAL: NCT02939989
Title: An Open-Label, Multicenter Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Combination With Sofosbuvir and Ribavirin in Chronic Hepatitis C (HCV) Infected Subjects Who Have Experienced Virologic Failure in AbbVie HCV Clinical Studies (MAGELLAN-3)
Brief Title: Efficacy and Safety of Glecaprevir (ABT-493)/Pibrentasvir (ABT 530) (GLE/PIB) in Combination With Sofosbuvir and Ribavirin in Participants With Hepatitis C Virus Who Did Not Respond to Treatment in a Previous AbbVie Clinical Study
Acronym: MAGELLAN-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15-942; 2016-002491-26 (EudraCT Number)
Expanded Access: NCT03123965 (Approved for marketing)
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Results first posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Hepatitis C Virus Infection
Keywords: Chronic Hepatitis C (HCV); HCV Genotype 1 (HCV GT1); HCV Genotype 2 (HCV GT2); HCV Genotype 3 (HCV GT3); HCV Genotype 4 (HCV GT4); HCV Genotype 5 (HCV GT5); HCV Genotype 6 (HCV GT6); Compensated Cirrhosis; Non-cirrhotics; Virologic failure
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — Sofosbuvir; glecaprevir and pibrentasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glecaprevir/Pibrentasvir + SOF + RBV for 12 weeks (Experimental): Participants without cirrhosis who had non-genotype 3 infection and were naïve to protease inhibitor (PI) and/or nonstructural viral protein 5A inhibitor (NS5Ai) prior to participation in AbbVie HCV parent study received daily treatment with glecaprevir/pibrentasvir (GLE/PIB) 300 mg/120 mg plus sofosbuvir (SOF) 400 mg plus twice-daily weight-based ribavirin (RBV) 600 mg - 1200 mg daily total for 12 weeks.
  Interventions: Drug: Sofosbuvir; Drug: Glecaprevir/Pibrentasvir; Drug: Ribavirin
- Glecaprevir/Pibrentasvir + SOF + RBV for 16 weeks (Experimental): Participants with genotype 3, and/or compensated cirrhosis, and/or experience with PI and/or NS5Ai prior to participation in Abbvie HCV parent study received daily treatment with GLE/PIB 300 mg/120 mg plus SOF 400 mg plus twice-daily weight-based RBV 600 mg - 1200 mg daily total for 16 weeks.
  Interventions: Drug: Sofosbuvir; Drug: Glecaprevir/Pibrentasvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Sofosbuvir — Tablet for oral administration
  Other Names: SOVALDI
Drug: Glecaprevir/Pibrentasvir — Coformulated tablet for oral administration
  Other Names: ABT-493/ABT-530; MAVYRET; MAVIRET
Drug: Ribavirin — Tablet for oral administration

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of co-administration of glecaprevir (ABT-493)/pibrentasvir (ABT 530) plus sofosbuvir (SOF) plus ribavirin (RBV) in hepatitis C virus (HCV) genotype (GT) 1 - 6-infected participants (including non-cirrhotic, or cirrhotic with compensated cirrhosis participants) who had experienced virologic failure in an AbbVie parent clinical study.

DETAILED DESCRIPTION:
This study enrolled HCV infected adults who had experienced virologic failure following treatment with glecaprevir/pibrentasvir or paritaprevir/ritonavir/ombitasvir + dasabuvir (DSV) (3D) or paritaprevir/ritonavir/ombitasvir (2D) regimens in one of the following AbbVie hepatitis C virus parent studies:

* M13-594 (NCT02640157)
* M13-596 (NCT02692703)
* M14-172 (NCT02642432)
* M14-242 (NCT02493855)
* M14-868 (NCT02243293)
* M15-410 (NCT02446717)
* M15-592 (NCT03222583)
* M16-126 (NCT02966795)
* M16-135 (NCT03089944)

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects must be adults (18 years of age or older) or adolescents (12 to less than 18 years of age weighing at least 35 kg).
* Subject must have experienced virologic failure during or after treatment with ABT-493/ABT-530 in an AbbVie HCV parent study. Subjects who have experienced virologic failure during or after receiving ombitasvir/paritaprevir/r + dasabuvir (3D), or ombitasvir/paritaprevir/r (2D) in an AbbVie HCV parent study may be enrolled at AbbVie's discretion. Treatment in the parent study must have been completed or discontinued at least 1 month prior to the Screening Visit.
* Subjects must be able to understand and adhere to the study visit schedule and all other protocol requirements.
* Cirrhotic subjects must have compensated cirrhosis, (Child-Pugh score of ≤ 6) at Screening and no current or past evidence of Child-Pugh B or C Classification or no clinical history of liver decompensation, including ascites noted on physical exam, hepatic encephalopathy or esophageal variceal bleeding.
* Cirrhotic subjects must have absence of hepatocellular carcinoma (HCC) as indicated by a negative ultrasound (US), computed tomography (CT) scan or magnetic resonance imaging (MRI) within 3 months prior to Screening or a negative US at Screening.

Exclusion Criteria:

* History of severe, life-threatening or other clinically significant sensitivity to any study drug or drug component.
* Female subject who is pregnant, breastfeeding or is considering becoming pregnant during the study or for 4 months after the last dose of study drug, or as directed per the local RBV label, whichever is more restrictive.
* Recent (within 6 months prior to study drug administration) history of drug or alcohol abuse that could preclude adherence to the protocol in the opinion of the investigator.
* Positive test result at Screening for hepatitis B surface antigen (HBsAg).
* Screening laboratory analyses showing calculated creatinine clearance < 30 mL/min.
* Discontinuation from the AbbVie HCV parent study for reasons other than virologic failure (e.g., non-adherence, lost to follow-up, and/or the occurrence of an adverse event).
* Receipt of any HCV treatment after failing the treatment regimen in the AbbVie HCV parent study.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (26):
- United States (8):
  - Digestive Health Specialists of the Southeast /ID# 155719, Dothan, Alabama
  - Ruane Clinical Research Group /ID# 155714, Los Angeles, California
  - Digestive Disease Associates - Baltimore /ID# 155713, Baltimore, Maryland
  - Henry Ford Health System /ID# 155720, Detroit, Michigan
  - University of Buffalo /ID# 155721, Buffalo, New York
  - Carolinas Center For Liver Dis /ID# 155731, Statesville, North Carolina
  - Gastro One /ID# 155729, Germantown, Tennessee
  - TX Liver Inst, Americ Res Corp /ID# 157881, San Antonio, Texas
- Australia (2):
  - Royal Brisbane and Women's Hospital /ID# 200944, Herston, Queensland
  - The Royal Melbourne Hospital /ID# 155727, Parkville, Victoria
- University of Calgary /ID# 155726, Calgary, Alberta, Canada
- China (4):
  - Beijing Di Tan Hospital, Capital Medical University /ID# 218496, Beijing
  - West China Hospital, Sichuan University /ID# 217613, Chengdu
  - The First Hospital Affiliated to AMU (Southwest Hospital) /ID# 218494, Chongqing
  - Mengchao Hepatobiliary Hospital of Fujian Medical University /ID# 218495, Fuzhou
- Germany (2):
  - Zentru fur HIV und Heaptogastroenterologie /ID# 155592, Düsseldorf, North Rhine-Westphalia
  - Asklepios Klinik St. Georg /ID# 155733, Hamburg
- New Zealand (3):
  - Auckland City Hospital /ID# 200945, Grafton, Auckland
  - Dunedin Hospital /ID# 155591, Otago, Otago
  - Waikato Hospital /ID# 155728, Hamilton, Waikato Region
- Medical Company Hepatolog /ID# 214314, Samara, Samara Oblast, Russia
- Samsung Medical Center /ID# 214844, Seoul, South Korea
- Hospital Universitario Puerta de Hierro, Majadahonda /ID# 155734, Majadahonda, Madrid, Spain
- Duplicate_Karolinska Univ Sjukhuset /ID# 155735, Solna, Sweden
- Inselspital, Universitätsspital Bern /ID# 155716, Bern, Switzerland
- Duplicate_Imperial College Healthcare NHS Trust /ID# 155718, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Background] Wyles D, Weiland O, Yao B, Weilert F, Dufour JF, Gordon SC, Stoehr A, Brown A, Mauss S, Zhang Z, Pilot-Matias T, Rodrigues L Jr, Mensa FJ, Poordad F. Retreatment of patients who failed glecaprevir/pibrentasvir treatment for hepatitis C virus infection. J Hepatol. 2019 May;70(5):1019-1023. doi: 10.1016/j.jhep.2019.01.031. Epub 2019 Mar 8. No abstract available. PMID 30857780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with hepatitis C virus (HCV) genotypes (GT) 1-6 infection who had virologic failure while participating in an AbbVie HCV Parent Study were enrolled at 26 sites in 12 countries.
Pre-assignment Details: Participants were allocated to 1 of 2 treatment arms based on HCV GT, cirrhosis status, and treatment experience with protease inhibitor (PI) and/or nonstructural viral protein 5A protease inhibitor (NS5Ai)-containing regimens prior to enrolling in the AbbVie HCV Parent Study.
Period: Overall Study
Arm/Group | Glecaprevir/Pibrentasvir + SOF + RBV for 12 Weeks | Glecaprevir/Pibrentasvir + SOF + RBV for 16 Weeks
Started | 5 | 28
Completed | 5 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Glecaprevir/Pibrentasvir + SOF + RBV for 12 Weeks: Participants without cirrhosis who had non-genotype 3 infection and were naïve to PI and/or NS5Ai prior to participation in AbbVie HCV parent study received daily treatment with GLE/PIB 300 mg/120 mg plus SOF 400 mg plus twice-daily weight-based RBV 600 mg - 1200 mg daily total for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Glecaprevir/Pibrentasvir + SOF + RBV for 12 Weeks | Glecaprevir/Pibrentasvir + SOF + RBV for 16 Weeks | Total
Number analyzed (Participants) | 5 | 28 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (8.08) | 54.3 (9.35) | 55.1 (9.25)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 3 | 23 | 26
  ≥ 65 years | 2 | 5 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 4 | 24 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 5 | 26 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 22 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
HCV Genotype [Count of Participants; unit: Participants]
  Genotype 1 | 1 | 7 | 8
  Genotype 2 | 4 | 0 | 4
  Genotype 3 | 0 | 19 | 19
  Genotype 4 | 0 | 1 | 1
  Genotype 5 | 0 | 0 | 0
  Genotype 6 | 0 | 1 | 1
AbbVie HCV Parent Study [Count of Participants; unit: Participants]
  M13-594 (NCT02640157) | 0 | 9 | 9
  M13-596 (NCT02692703) | 0 | 1 | 1
  M14-172 (NCT02642432) | 0 | 1 | 1
  M14-242 (NCT02493855) | 1 | 0 | 1
  M14-868 (NCT02243293) | 2 | 6 | 8
  M15-410 (NCT02446717) | 0 | 6 | 6
  M15-592 (NCT03222583) | 2 | 3 | 5
  M16-126 (NCT02966795) | 0 | 1 | 1
  M16-135 (NCT03089944) | 0 | 1 | 1
Treatment Regimen Received in AbbVie HCV Parent Study [Count of Participants; unit: Participants] — GLE/PIB = glecaprevir/pibrentasvir; OBV/PTV/RTV + DSV + RBV = ombitasvir/paritaprevir/ritonavir + dasabuvir (VIEKIRAX and EXVIERA) + ribavirin
  Participants
    GLE/PIB | 4 | 28 | 32
    OBV/PTV/RTV + DSV + RBV | 1 | 0 | 1
Treatment Response for AbbVie HCV Parent Study [Count of Participants; unit: Participants] — On-treatment non-responder: HCV RNA ≥ 15 IU/ml at end of treatment with at least 6 weeks of treatment.
  Breakthrough: Confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < 15 IU/ml during the Treatment Period; or confirmed increase from nadir in HCV RNA (two consecutive HCV RNA measurements > 1 log10 IU/mL above nadir) at any time during the Treatment Period.
  Relapse: Confirmed HCV RNA ≥ 15 IU/ml between end of treatment and the last HCV RNA measurement collected in the Post-Treatment Period if HCV RNA < 15 IU/ml at Final Treatment Visit and treatment was completed.
  Participants
    On-treatment non-responder | 0 | 10 | 10
    Breakthrough | 0 | 0 | 0
    Post-treatment relapse | 5 | 18 | 23
HCV Ribonucleic Acid (RNA) Level [Mean (Standard Deviation); unit: log10 IU/mL] | 6.79 (0.217) | 6.23 (0.958) | 6.32 (0.907)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification (LLOQ; 15 IU/mL) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug, Week 24 or Week 28 depending on the treatment regimen.
Population: Intention-to-treat (ITT) population, which included all participants who received at least 1 dose of study drug. A backward imputation method was used to impute missing responses. Participants with missing data after backward imputation were counted as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Total: Participants received daily treatment with GLE/PIB 300 mg/120 mg plus SOF 400 mg plus twice-daily weight-based RBV 600 mg - 1200 mg daily total for 12 or 16 weeks.
Arm/Group | Glecaprevir/Pibrentasvir + SOF + RBV for 12 Weeks | Glecaprevir/Pibrentasvir + SOF + RBV for 16 Weeks | Total
Number analyzed (Participants) | 5 | 28 | 33
percentage of participants | 100 [56.6 to 100.0] | 96.4 [82.3 to 99.4] | 97.0 [84.7 to 99.5]

2. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as meeting one of the following:
  * confirmed increase from nadir in HCV RNA (two consecutive HCV RNA measurements > 1 log10 IU/mL above nadir) at any time point during the treatment period; or
  * confirmed HCV RNA greater than or equal to 100 IU/mL after HCV RNA < 15 IU/mL during the treatment period, or
  * HCV RNA ≥ 15 IU/mL at end of treatment with at least 6 weeks of treatment.
Time Frame: 12 or 16 weeks depending on the treatment regimen
Population: Intention-to-treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir + SOF + RBV for 12 Weeks | Glecaprevir/Pibrentasvir + SOF + RBV for 16 Weeks | Total
Number analyzed (Participants) | 5 | 28 | 33
percentage of participants | 0 [0.0 to 43.4] | 0 [0.0 to 12.1] | 0 [0.0 to 10.4]

3. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA greater than or equal to 15 IU/mL between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < 15 IU/mL at the end of treatment, and had post-treatment HCV RNA data; participants who had been shown to be re-infected were not considered to have relapsed.
Time Frame: From the end of treatment (Week 12 or 16) through 12 weeks after the last dose of study drug (Weeks 24 or 28 depending on the treatment regimen).
Population: Intention-to-treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir + SOF + RBV for 12 Weeks | Glecaprevir/Pibrentasvir + SOF + RBV for 16 Weeks | Total
Number analyzed (Participants) | 5 | 28 | 33
percentage of participants | 0 [0.0 to 43.4] | 3.6 [0.6 to 17.7] | 3.0 [0.5 to 15.3]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose; up to 20 weeks.
Groups:
- GLE/PIB + SOF + RBV for 12 Weeks: Participants without cirrhosis who had non-genotype 3 infection and were naïve to PI and NS5Ai prior to participation in AbbVie HCV parent study received daily treatment with GLE/PIB 300 mg/120 mg plus SOF 400 mg plus twice-daily weight-based RBV 600 mg - 1200 mg daily total for 12 weeks.
- GLE/PIB + SOF + RBV for 16 Weeks: Participants with genotype 3, and/or compensated cirrhosis, and/or experience with PI and/or NS5Ai prior to participation in Abbvie HCV parent study received daily treatment with GLE/PIB 300 mg/120 mg plus SOF 400 mg plus twice-daily weight-based RBV 600 mg - 1200 mg daily total for 16 weeks.
Arm/Group | GLE/PIB + SOF + RBV for 12 Weeks | GLE/PIB + SOF + RBV for 16 Weeks | Total
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/28 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/5 | 2/28 | 3/33
Other Adverse Events (participants affected / at risk) | 5/5 | 21/28 | 26/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLE/PIB + SOF + RBV for 12 Weeks (N=5) | GLE/PIB + SOF + RBV for 16 Weeks (N=28) | Total (N=33)
CHRONIC GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLE/PIB + SOF + RBV for 12 Weeks (N=5) | GLE/PIB + SOF + RBV for 16 Weeks (N=28) | Total (N=33)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
ASTHENIA (General disorders) | 0 (0) | 3 (3) | 3 (3)
FATIGUE (General disorders) | 1 (1) | 3 (3) | 4 (4)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0) | 1 (1)
MALAISE (General disorders) | 1 (1) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 4 (4) | 4 (4)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 1 (1) | 2 (2)
HAEMATOCRIT DECREASED (Investigations) | 1 (1) | 0 (0) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 1 (1) | 2 (2)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 1 (1)
MEAN CELL VOLUME INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1)
RED BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 1 (1)
WEIGHT DECREASED (Investigations) | 1 (1) | 1 (1) | 2 (2)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 4 (4) | 5 (5)
HEADACHE (Nervous system disorders) | 1 (1) | 5 (6) | 6 (7)
INSOMNIA (Psychiatric disorders) | 1 (1) | 3 (3) | 4 (4)
IRRITABILITY (Psychiatric disorders) | 0 (0) | 4 (4) | 4 (4)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (3)
LARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (2) | 6 (6) | 7 (8)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT02939989/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT02939989/SAP_001.pdf